CLINICAL TRIAL: NCT03138356
Title: A Randomized, Single-dose, Open-label, Single-center, Crossover Study to Assess the Fed- and Fasted State Bioequivalence of Fixed-Dose Combination Tablets of Saxagliptin / Dapagliflozin / Metformin XR and Dapagliflozin / Metformin XR Relative to Individual Components in Healthy Subjects
Brief Title: Bioequivalence Study of Combination Tablets of Saxagliptin / Dapagliflozin / Metformin XR (Extended-release) and Dapagliflozin / Metformin XR Relative to Individual Components in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: D168AC00002
Record Dates: First submitted 2017-04-21; First posted 2017-05-03 (Actual); Last update posted 2017-12-07 (Actual); Status verified 2017-12

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Type 2 diabetes mellitus, saxagliptin, dapagliflozin, metformin XR, fixed-dose combination, healthy subjects, crossover, cohorts.
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — saxagliptin; dapagliflozin; Tablets; Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (9):
- Cohort 1 Treatment A (Experimental): Single-dose of saxagliptin (2.5 mg), dapagliflozin (5 mg), metformin (1000 mg) XR (Extended-release) FDC (Fixed-dose combination) tablet administered orally under fasted condition. Within each cohort, subjects will be randomized to 1 of 6 treatment sequences, each subject will receive 3 single-dose treatments in either a fasted or fed-state.
  The treatment sequences are (ABC), (ACB), (BAC), (BCA), (CAB) or (CBA).
  Interventions: Drug: 2.5 mg saxagliptin / 5 mg dapagliflozin / 1000 mg metformin XR FDC tablet
- Cohort 1 Treatment B (Experimental): Single-dose of saxagliptin (2.5 mg), dapagliflozin (5 mg), metformin (850 mg) XR FDC tablet, administered orally under fasted condition. Within each cohort, subjects will be randomized to 1 of 6 treatment sequences, each subject will receive 3 single-dose treatments in either a fasted or fed-state.
  The treatment sequences are (ABC), (ACB), (BAC), (BCA), (CAB) or (CBA).
  Interventions: Drug: 2.5 mg saxagliptin / 5 mg dapagliflozin / 850 mg metformin XR FDC tablet
- Cohort 1 Treatment C (Reference product) (Active Comparator): Single-dose of Onglyza® (2.5 mg saxagliptin), Forxiga® (5 mg dapagliflozin) and Glucophage XR® (2 x 500 mg metformin XR) co-administered under fasted condition. Within each cohort, subjects will be randomized to 1 of 6 treatment sequences, each subject will receive 3 single-dose treatments in either a fasted or fed-state.
  The treatment sequences are (ABC), (ACB), (BAC), (BCA), (CAB) or (CBA).
  Interventions: Drug: 2.5 mg ONGLYZA® (saxagliptin) tablet; Drug: 5 mg Forxiga® (dapagliflozin) tablet; Drug: 500 mg Glucophage XR®
- Cohort 2 Treatment D (Experimental): Single-dose of saxagliptin (2.5 mg), dapagliflozin (5 mg), metformin (1000 mg) XR FDC tablet administered orally under fed condition. Within each cohort, subjects will be randomized to 1 of 6 treatment sequences, each subject will receive 3 single-dose treatments in either a fasted or fed-state
  The treatment sequences are (DEF), (DFE), (EDF), (EFD), (FDE) or (FED).
  Interventions: Drug: 2.5 mg saxagliptin / 5 mg dapagliflozin / 1000 mg metformin XR FDC tablet
- Cohort 2 Treatment E (Experimental): Single-dose of saxagliptin (2.5 mg), dapagliflozin (5 mg), metformin (850 mg) XR FDC tablet, administered orally under fed condition. Within each cohort, subjects will be randomized to 1 of 6 treatment sequences, each subject will receive 3 single-dose treatments in either a fasted or fed-state.
  The treatment sequences are (DEF), (DFE), (EDF), (EFD), (FDE) or (FED).
  Interventions: Drug: 2.5 mg saxagliptin / 5 mg dapagliflozin / 850 mg metformin XR FDC tablet
- Cohort 2 Treatment F (Reference Product) (Active Comparator): Single-dose of Onglyza® (2.5 mg saxagliptin), Forxiga® (5 mg dapagliflozin) and Glucophage XR® (2 x 500 mg metformin) co-administered under fed condition. Within each cohort, subjects will be randomized to 1 of 6 treatment sequences, each subject will receive 3 single-dose treatments in either a fasted or fed-state.
  The treatment sequences are (DEF), (DFE), (EDF), (EFD), (FDE) or (FED).
  Interventions: Drug: 2.5 mg ONGLYZA® (saxagliptin) tablet; Drug: 5 mg Forxiga® (dapagliflozin) tablet; Drug: 500 mg Glucophage XR®
- Cohort 3 Treatment G (Experimental): Single-dose dapagliflozin (5 mg) / metformin (1000 mg) XR FDC tablet administered orally under fed condition. Within each cohort, subjects will be randomized to 1 of 6 treatment sequences, each subject will receive 3 single-dose treatments in either a fasted or fed-state.
  The treatment sequences are (GHI), (GIH), (HGI), (HIG), (IHG) or (IGH).
  Interventions: Drug: 5 mg dapagliflozin / 1000 mg metformin XR FDC
- Cohort 3 Treatment H (Experimental): Single-dose dapagliflozin (5 mg) / metformin (850 mg) XR FDC tablet administered orally under fed condition. Within each cohort, subjects will be randomized to 1 of 6 treatment sequences, each subject will receive 3 single-dose treatments in either a fasted or fed-state.
  The treatment sequences are (GHI), (GIH), (HGI), (HIG), (IHG) or (IGH).
  Interventions: Drug: 5 mg dapagliflozin / 850 mg metformin XR FDC
- Cohort 3 Treatment I (Reference Product) (Active Comparator): Single-dose Forxiga® (5 mg dapagliflozin) and Glucophage XR® (2 x 500 mg metformin) co-administered under fed condition. Within each cohort, subjects will be randomized to 1 of 6 treatment sequences, each subject will receive 3 single-dose treatments in either a fasted or fed-state.
  The treatment sequences are (GHI), (GIH), (HGI), (HIG), (IHG) or (IGH).
  Interventions: Drug: 5 mg Forxiga® (dapagliflozin) tablet; Drug: 500 mg Glucophage XR®

INTERVENTIONS:
Drug: 2.5 mg saxagliptin / 5 mg dapagliflozin / 850 mg metformin XR FDC tablet — Used in Treatment B and Treatment E.
  Arms: Cohort 1 Treatment B; Cohort 2 Treatment E
Drug: 2.5 mg saxagliptin / 5 mg dapagliflozin / 1000 mg metformin XR FDC tablet — Used in Treatment A and Treatment D.
  Arms: Cohort 1 Treatment A; Cohort 2 Treatment D
Drug: 5 mg dapagliflozin / 850 mg metformin XR FDC — Used in Treatment H.
  Arms: Cohort 3 Treatment H
Drug: 5 mg dapagliflozin / 1000 mg metformin XR FDC — Used in Treatment G.
  Arms: Cohort 3 Treatment G
Drug: 2.5 mg ONGLYZA® (saxagliptin) tablet — Used in treatments C and F.
  Arms: Cohort 1 Treatment C (Reference product); Cohort 2 Treatment F (Reference Product)
Drug: 5 mg Forxiga® (dapagliflozin) tablet — Used in treatments C, F and I.
  Arms: Cohort 1 Treatment C (Reference product); Cohort 2 Treatment F (Reference Product); Cohort 3 Treatment I (Reference Product)
Drug: 500 mg Glucophage XR® — Used in treatments C, F and I.
  Arms: Cohort 1 Treatment C (Reference product); Cohort 2 Treatment F (Reference Product); Cohort 3 Treatment I (Reference Product)

SUMMARY:
In this integrated, Phase I study, the safety, tolerability, food effect, and pharmacokinetic (PK) properties of Fixed-Dose Combination Tablets of Saxagliptin / Dapagliflozin / Metformin XR and Dapagliflozin / Metformin XR Relative to Individual Components in Healthy Subjects will be investigated.

DETAILED DESCRIPTION:
This study will be an open-label, randomized, 3-period, 3-treatment, single-dose crossover study in healthy subjects (males and females), performed at a single study center, conducted in 3 cohorts. A total of 126 healthy male or female subjects (3 cohorts of 42 subjects each [each cohort consisting of 3 treatments]) will be randomized in this study to ensure that at least 108 subjects (36 in each cohort) are evaluable. Each subject will receive 3 single-dose treatments, and each treatment will be administered within 1 of the 3 successive treatment periods. Within each cohort, subjects will be randomized to 1 of 6 treatment sequences with 7 subjects prescribing the ordered sequence of 3 administered treatments in each treatment sequence, and will receive the IMPs in either a fasted or fed-state according to the assigned treatment. For fed-state cohorts, all doses of study drug will be administered to subjects after consuming a standard meal (light fat, low calorie) in the morning. Subjects will start consuming the meal 30 minutes prior to the dose and will finish the meal within 25 minutes. Dosing will then start after 30 minutes after the start of the meal. Subjects in the fasted state cohort will be fasted overnight (at least 10 hours) before dosing

The study will comprise:

* A Screening period of maximum 28 days;
* Three treatment periods during which subjects will be resident in the Unit from the day before dosing with the IMP (Day -1) until at least 72 hours after dosing; discharged on the morning of Day 4; and
* A final Follow-up Visit within 5 to 7 days after the last administration of the IMP.

There will be a minimum washout period of 7 to 14 days between each dose administration

ELIGIBILITY:
Inclusion Criteria:

* For inclusion in the study subjects should fulfill the following criteria:

  1. Provision of signed and dated, written informed consent prior to any study specific procedures.
  2. Healthy male and/or female subjects aged 18 to 55 years with suitable veins for cannulation or repeated venipuncture.
  3. Female subject must either:

3.1. Be of non-childbearing potential:

* Must have a negative serum pregnancy test (minimum sensitivity 25 IU/L or equivalent units of human chorionic gonadotropin) at Screening and negative urine pregnancy test within 24 hours prior to first IMP administration.
* Documentation of irreversible surgical sterilization by hysterectomy, bilateral oophorectomy or bilateral salpingectomy but not tubal ligation. 3.2. Or, if of childbearing potential:
* Must have a negative serum pregnancy test (minimum sensitivity 25 IU/L or equivalent units of human chorionic gonadotropin) at Screening and within 24 hours prior to first IMP administration.
* Must not be nursing (breastfeeding).
* If heterosexually active, agree to consistently use a highly effective method of contraception to avoid pregnancy, from at least 4 weeks prior to dosing and throughout the study and for up to 90 days after the last dose of IMP. 4. Sexually active fertile male subjects must use effective birth control for the entire study and 90 days after the last dose of IMP if their partners are women of childbearing potential. 5. Have a body mass index (BMI) between 18 and 32 kg/m2 inclusive and weigh at least 50 kg and no more than 100 kg inclusive.

Exclusion Criteria:

* Subjects will not enter the study if any of the following exclusion criteria are fulfilled:

  1. History of any clinically significant disease or disorder which, in the opinion of the PI, may either put the volunteer at risk because of participation in the study, or influence the results or the volunteer's ability to participate in the study.
  2. Current or recent (within 3 months of first IMP dosing) gastrointestinal disease that may impact drug absorption and affect the PK of the study drugs. Additionally, any gastrointestinal surgery (e.g., partial gastrectomy, pyloroplasty) including cholecystectomy that may impact drug absorption.
  3. Any major surgery, as determined by the investigator, within 4 weeks of first IMP dosing.
  4. Donation of > 400 mL of blood within 8 weeks or donation of plasma (except at the Screening Visit) within 4 weeks of first IMP dosing.
  5. Blood transfusion within 4 weeks of first IMP dosing.
  6. Inability to tolerate oral medication.
  7. Inability to tolerate venipuncture or inadequate venous access as determined by the investigator.
  8. Recent (within 6 months of first IMP dosing) drug or alcohol abuse as defined in the Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition (DSM-IV), Diagnostic Criteria for Drug and Alcohol Abuse.
  9. Subjects who drink more than 3 cups of coffee or other caffeinecontaining products a day, or 5 cups of tea a day.
  10. Use of tobacco-containing or nicotine-containing products (including but not limited to cigarettes, pipes, cigars, chewing tobacco, nicotine patches, nicotine lozenges, or nicotine gum) within 6 months prior to first check-in (Day -1, Treatment Period 1), or a positive nicotine test (i.e., cotinine) at Screening and/or check-in.
  11. History of diabetes mellitus.
  12. History of heart failure.
  13. History of chronic or recurrent urinary tract infection (defined as 3 occurrences per year)
  14. Recent vulvovaginal mycotic infection (within 2 months prior to first IMP dosing).
  15. Any other sound medical, psychiatric and/or social reason as determined by the investigator.
  16. Any clinically significant illness, medical/surgical procedure, or trauma within 4 weeks of Screening.
  17. Any positive result on screening for serum hepatitis B surface antigen, hepatitis C antibody, and human immunodeficiency virus (HIV) antibody.
  18. Has received another new chemical entity (defined as a compound which has not been approved for marketing) within 3 months of the first administration of IMP in this study. The period of exclusion begins 3 months after the final dose or one month after the last visit whichever is the longest. Note: subjects consented and screened, but not randomized in this study or a previous Phase1 study, are not excluded.
  19. History of severe allergy/hypersensitivity or ongoing allergy/hypersensitivity, as judged by the PI or history of hypersensitivity to drugs with a similar chemical structure or class to saxagliptin, dapagliflozin and metformin.
  20. Positive screen for drugs of abuse or cotinine at Screening or on first admission to the study center or positive screen for alcohol on first admission to the study center
  21. Use of saxagliptin, dapagliflozin and/or metformin within 3 months prior to the first administration of IMP.
  22. Use of any prescription drugs or OTC acid controllers within 4 weeks prior to the first administration of IMP except medication cleared by the medical monitor.
  23. Use of drugs with enzyme-inducing properties such as St John's Wort within 3 weeks prior to the first administration of IMP.
  24. Use of any prescribed or non-prescribed medication including analgesics (other than paracetamol/acetaminophen), herbal remedies, megadose vitamins (intake of 20 to 600 times the recommended daily dose) and minerals during the 2 weeks prior to the first administration of IMP or longer if the medication has a long half-life. Note: Hormonal replacement therapy is not allowed.
  25. Involvement of any AstraZeneca, PAREXEL or study site employee or their close relatives.
  26. Vulnerable subjects, e.g., kept in detention, protected adults under guardianship, trusteeship, or committed to an institution by governmental or juridical order.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 126 (Actual)
Dates: Start 2017-05-25 (Actual); Primary Completion 2017-11-28 (Actual); Study Completion 2017-11-28 (Actual)

PRIMARY OUTCOMES:
PK assessment: AUC (Area under plasma concentration-time curve from time zero to infinity) | At Pre-dose, 0.25, 0.5, 1, 1.5, 2,3,4,6,8,12, 18, 24,36, 48, 60 and 72 hours (Days 1 to 4)
  To measure the PK exposure for saxagliptin, 5-hydroxy saxagliptin (where applicable), dapagliflozin and metformin using plasma concentrations in subjects following IMP administration.
PK assessment: AUC0-t (Area under the plasma concentration-time curve from time zero to time of last quantifiable concentration) | At Pre-dose, 0.25, 0.5, 1, 1.5, 2,3,4,6,8,12, 18, 24,36, 48, 60 and 72 hours (Days 1 to 4)
  To measure the PK exposure for saxagliptin, 5-hydroxy saxagliptin (where applicable), dapagliflozin and metformin using plasma concentrations in subjects following IMP administration.
PK assessment: Cmax (Maximum observed plasma concentration) | At Pre-dose, 0.25, 0.5, 1, 1.5, 2,3,4,6,8,12, 18, 24,36, 48, 60 and 72 hours (Days 1 to 4)
  To measure the PK exposure for saxagliptin, 5-hydroxy saxagliptin (where applicable), dapagliflozin and metformin using plasma concentrations in subjects following IMP administration.

SECONDARY OUTCOMES:
Secondary PK parameter: tmax (Time to reach maximum observed plasma concentration) | At Pre-dose, 0.25, 0.5, 1, 1.5, 2,3,4,6,8,12, 18, 24,36, 48, 60 and 72 hours (Days 1 to 4)
  To measure the PK exposure for saxagliptin, 5-hydroxy saxagliptin (where applicable), dapagliflozin and metformin using plasma concentrations in subjects following IMP administration.
Secondary PK parameter: t½,λz (Terminal elimination half-life) | At Pre-dose, 0.25, 0.5, 1, 1.5, 2,3,4,6,8,12, 18, 24,36, 48, 60 and 72 hours (Days 1 to 4)
  To measure the PK exposure for saxagliptin, 5-hydroxy saxagliptin (where applicable), dapagliflozin and metformin using plasma concentrations in subjects following IMP administration.
Secondary PK parameter: tlast (Time of last quantifiable plasma concentration) | At Pre-dose, 0.25, 0.5, 1, 1.5, 2,3,4,6,8,12, 18, 24,36, 48, 60 and 72 hours (Days 1 to 4)
  To measure the PK exposure for saxagliptin, 5-hydroxy saxagliptin (where applicable), dapagliflozin and metformin using plasma concentrations in subjects following IMP administration.
Secondary PK parameter: MRT (Mean residence time from zero to infinity (parent drug only)) | At Pre-dose, 0.25, 0.5, 1, 1.5, 2,3,4,6,8,12, 18, 24,36, 48, 60 and 72 hours (Days 1 to 4)
  To measure the PK exposure for saxagliptin, 5-hydroxy saxagliptin (where applicable), dapagliflozin and metformin using plasma concentrations in subjects following IMP administration.
Secondary PK parameter: λz (Terminal elimination rate constant) | At Pre-dose, 0.25, 0.5, 1, 1.5, 2,3,4,6,8,12, 18, 24,36, 48, 60 and 72 hours (Days 1 to 4)
  To measure the PK exposure for saxagliptin, 5-hydroxy saxagliptin (where applicable), dapagliflozin and metformin using plasma concentrations in subjects following IMP administration.
Secondary PK parameter: CL/F (Apparent total body clearance of drug from plasma after extravascular administration (parent drug only)) | At Pre-dose, 0.25, 0.5, 1, 1.5, 2,3,4,6,8,12, 18, 24,36, 48, 60 and 72 hours (Days 1 to 4)
  To measure the PK exposure for saxagliptin, 5-hydroxy saxagliptin (where applicable), dapagliflozin and metformin using plasma concentrations in subjects following IMP administration.
Secondary PK parameter: Vz/F (Apparent volume of distribution during terminal phase after extravascular administration (parent drug only)) | At Pre-dose, 0.25, 0.5, 1, 1.5, 2,3,4,6,8,12, 18, 24,36, 48, 60 and 72 hours (Days 1 to 4)
  To measure the PK exposure for saxagliptin, 5-hydroxy saxagliptin (where applicable), dapagliflozin and metformin using plasma concentrations in subjects following IMP administration.
Secondary PK parameters: AUC/D (Dose normalized AUC (metformin only)) | At Pre-dose, 0.25, 0.5, 1, 1.5, 2,3,4,6,8,12, 18, 24,36, 48, 60 and 72 hours (Days 1 to 4)
  To measure the PK exposure for saxagliptin, 5-hydroxy saxagliptin (where applicable), dapagliflozin and metformin using plasma concentrations in subjects following IMP administration.
Secondary PK parameter: AUC0-t/D (Dose normalized AUC0-t (metformin only)) | At Pre-dose, 0.25, 0.5, 1, 1.5, 2,3,4,6,8,12, 18, 24,36, 48, 60 and 72 hours (Days 1 to 4)
  To measure the PK exposure for saxagliptin, 5-hydroxy saxagliptin (where applicable), dapagliflozin and metformin using plasma concentrations in subjects following IMP administration.
Secondary PK parameter: Cmax/D (Dose normalized Cmax (metformin only)) | At Pre-dose, 0.25, 0.5, 1, 1.5, 2,3,4,6,8,12, 18, 24,36, 48, 60 and 72 hours (Days 1 to 4)
  To measure the PK exposure for saxagliptin, 5-hydroxy saxagliptin (where applicable), dapagliflozin and metformin using plasma concentrations in subjects following IMP administration.
Number of patients with Adverse Events (AEs) | At Day -1, Spontaneous plus Pre-dose, 3, 12, 24, and 48 hours post-dose (Days 1 to 4), 5 to 7 days post-final dose
  To assess the adverse events as a criteria of safety and tolerability variables.
Vital signs (systolic and diastolic blood pressure [BP]) | At Screening, Day -1, Pre-dose and 48 hours (Days 1 to 4), 5 to 7 days post-final dose]
  To assess the vital signs as a criteria of safety and tolerability variables.
Vital signs (pulse rate) | At Screening, Day -1, Pre-dose and 48 hours (Days 1 to 4), 5 to 7 days post-final dose]
  To assess the vital sign as a criteria of safety and tolerability variables.
Twelve-lead electrocardiograms (ECGs) | At Screening, 5 to 7 days post-final dose ]
  To assess the cardiovascular system functioning as a criteria of safety and tolerability variables.
Physical examination | At Screening, Day -1 (brief) , Day 4, 72 hours (brief) post-dose (Days 1 to 4), 5 to 7 days post-final dose ]
  To assess the physical conditions as a criteria of safety and tolerability variables.
Body weight | At Screening, Day -1, 5 to 7 days post-final dose ]
  To assess the body weight as a criteria of safety and tolerability variables.
Laboratory assessments (hematology, clinical chemistry and urinalysis) | At Screening, Day -1, Day 4 (72 hours post-dose), Post-study 5 to 7 days post-final dose
  To assess hematology, clinical chemistry and urinalysis as a criteria of safety and tolerability variables.

CONTACTS AND LOCATIONS:
Overall Officials: Pablo ForteSoto, MD, MSc, PhD, Principal Investigator — PAREXEL Early Phase Clinical Unit London
Locations (1):
- Research Site, Harrow, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided